CLINICAL TRIAL: NCT04434365
Title: The Study of Berberine Affecting Metabolism, Inflammation Status, Endothelial Function and Thrombotic Events in Patients With Coronary Artery Disease by Remodeling Gut Microbiota
Brief Title: Effect of Berberine for Endothelial Function and Intestinal Microflora in Patients With Coronary Artery Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBRCADGM2019; 2016-I2M-1-011 (Other Grant/Funding Number: CAMS Innovation Fund for Medical Sciences (CIFMS))
Record Dates: First submitted 2019-06-27; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Stable Coronary Artery Disease; Percutaneous Coronary Intervention
Keywords: Berberine; Gut microbiota; Endothelial function
MeSH Terms: interventions — Berberine; Aspirin; Clopidogrel; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: On the first day of the treatment period (Visit 1), eligible patients will be randomized into the Berberine Arm and the Control Arm.
  In the Berberine Arm, patients will receive berberine 200 mg twice daily for 4±1 weeks (Stage 1); then, 300 mg twice daily for 4±1 weeks (Stage 2); then, 400 mg twice daily for 4±1 weeks (Stage 3) in addition to standard treatment, including aspirin 100 mg once daily and clopidogrel 75 mg once daily for 12±1 weeks.
  In the Control Arm, patients will receive standard treatment, including aspirin 100 mg once daily and clopidogrel 75 mg once daily for 12±1 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Berberine+standard therapy Arm (Experimental): In the Berberine Arm, patients will receive berberine 100 mg twice daily for 4±1 weeks (Stage 1); then, 200 mg twice daily for 4±1 weeks (Stage 2); then, 300 mg twice daily for 4±1 weeks (Stage 3) in addition to standard treatment, including aspirin (100mg/day), clopidogrel (75mg/day), statins, the use of angiotensin-converting enzyme inhibitors or angiotensin receptor blockers, calcium channel blockers, beta-blockers, and/or antidiabetic therapy (including insulin or oral medication) was decided on an individual basis by the attending physician for 12±1 weeks.
  Interventions: Drug: Berberine; Drug: Aspirin; Drug: Clopidogrel; Drug: Statin
- Standard therapy Arm (Active Comparator): In the Control Arm, patients will receive standard treatment, including aspirin (100mg/day), clopidogrel (75mg/day), statins, the use of angiotensin-converting enzyme inhibitors or angiotensin receptor blockers, calcium channel blockers, beta-blockers, and/or antidiabetic therapy (including insulin or oral medication) was decided on an individual basis by the attending physician for 12±1 weeks.
  Interventions: Drug: Aspirin; Drug: Clopidogrel; Drug: Statin

INTERVENTIONS:
Drug: Berberine — Berberine 100 mg twice daily for 4±1 weeks (Stage 1); then, 200 mg twice daily for 4±1 weeks (Stage 2); then, 300 mg twice daily for 4 weeks (Stage 3).
  Other Names: Berberine Hydrochloride Tablets
  Arms: Berberine+standard therapy Arm
Drug: Aspirin — Aspirin 100 mg once daily for 12±1 weeks.
  Other Names: Aspirin Enteric-coated Tablets
Drug: Clopidogrel — Clopidogrel 75 mg once daily for 12±1 weeks.
  Other Names: Clopidogrel Hydrogen Sulphate Tablets; Plavix
Drug: Statin — Statins once daily for 12±1 weeks.
  Other Names: Atorvastatin; Rosuvastatin

SUMMARY:
The purpose of this study is to conduct a single-center, randomized, open-label, controlled, dose-escalating, parallel-group study, evaluating the effects and change of endothelial function and gut microbiota after berberine administration in patients with stable coronary artery disease who are at > 8 but ≤ 40 weeks after elective percutaneous coronary intervention

DETAILED DESCRIPTION:
In the present study, about 48 patients with stable coronary artery disease who are at > 8 but ≤ 40 weeks after elective percutaneous coronary intervention. The total study duration is expected to be approximately 14 weeks per patient, including a screening period, a 12±1 week treatment period, Randomization was computer generated. After screening, eligible subjects will be randomly assigned into one of the following two groups: Berberine+therapy Arm or Standard therapy Arm. The primary objective is to determine whether a combination of berberine and coronary artery disease standard therapy is preferable to either berberine alone or standard therapy alone.

The visit schedule will be as follows:

Visit 1: Day -7 to Day -1, Screening/Enrolment; Visit 2: Day 1, Randomization/First dose; Visit 3: Week 4±1, Dose adjustment 1, BBR (100mg, tid); Visit 4: Week 8±1, Dose adjustment 2, BBR (200mg, tid); Visit 5: Week 12±1, End of Treatment (EOT) /Last dose, BBR (300mg, tid); Safety visit.

We perform cross-sectional comparisons between the two arms and longitudinal comparisons within each arm to evaluate the indicators as follows:

1. . Endothelial function, as measured by Flow mediated dilation (FMD) from baseline to 12-week follow-up;
2. . Gut microbiota, as sequenced by metagenomic sequencing from baseline to 12-week follow-up.

Blood and feces samples will be collected before and after treatment. Flow mediated dilation (FMD), HbA1C, fasting plasma glucose (FPG), lipids and cholesterol level, inflammatory factors, amino acids, bile acids and other metabolic related components and parameters will be measured. Furthermore, the change of gut microbiota will be evaluated too.

ELIGIBILITY:
Inclusion Criteria:

Patients with stable coronary artery disease undergo elective PCI >8 weeks, but ≤40 weeks

Exclusion Criteria:

1. Planned coronary revascularization, including PCI and coronary artery bypass graft (CABG) during the study period.
2. Subjects with uncontrolled high blood pressure
3. Recent (within 4 weeks) dose adjustment of any standard therapy agents
4. Recent (within 4 weeks) use of berberine
5. History of intolerance to berberine.
6. Cr>1.5mg/dL; ALT level exceeds the upper limit of 3 times
7. Heart failure or LVEF <50%
8. Uncontrolled arrhythmia
9. Pregnancy or lactation
10. Malignant tumor or life expectancy is less than half a year
11. Subjects who can not complete the follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Endothelial function measured by Flow mediated dilation (FMD) | On the baseline, 4th, 8th, 12th week of treatment
  Flow-mediated vasodilation measurement in the brachial artery was performed with subjects in the supine position for the evaluation of endothelial function. All imaging was performed by a single, highly skilled sonographer who was unaware of the study assignment.brachial artery diameter was imaged with a 5-12-MHz linear array transducer ultrasound system at a location 3 to 7 cm above the right elbow. The brachial artery diameters at baseline (D0) and after reactive hyperemia (D1) and sublingual nitroglycerine (D2) were recorded. The flow-mediated vasodilation [(D1-D0)/D0×100%] was used as a measure of endothelium-dependent vasodilation.
Gut microbiome | On the baseline, 4th, 8th, 12th week of treatment
  At baseline, we evaluate the bacterial diversity, different species, different genes, and different metabolic pathways in the BBR+Standard therapy group and the Standard therapy group . In addition, we mainly focused on α and β diversity variation in the remaining 3 visits of BBR+Standard therapy subjucts. Taxonomy alteration and bacterial metabolic pathways after BBR treatment were also observed.
Fecal metabolomics profile measurement | On the baseline, 4th, 8th, 12th week of treatment
  In aid of LC/MS and GC/MS technique, we will measure the metabolomics molecular profile in fecal samples at baseline, 4th, 8th, 12th week. We aimed to detect the profile of short chain fatty acids including Acetic acid, Propanoic acid, Isobutyric acid, Butyric acid, Ethylmethylacetic acid, Isovaleric acid, Valeric acid, 2-methylvaleric acid, 3-methylvaleric acid, 4-methylvaleric acid, Hexanoic acid-SCFA and 3_Hydroxyisovaleric acid.

SECONDARY OUTCOMES:
Blood lipid levels | On the baseline, 4th, 8th, 12th week of treatment
  Total cholesterol (mmol/L), Triglyceride (mmol/L), HDL-C (mmol/L), LDL-C (mmol/L), Free fatty acids (umol/L), ApoA1(g/L), ApoB (g/L), Lp(a) (mg/L).
Inflammatory factor levels | On the 12th week of treatment
  hs-CRP (mg/L), IL-1b (pg/mL), IL-6 (pg/mL), IL-18 (pg/mL), TNF-a (pg/mL), IFN-r (pg/mL), IL-10 (pg/mL).
Blood glucose levels | On the baseline, 4th, 8th, 12th week of treatment
  Fasting glucose level (mmol/L), 2-hour postprandial glucose levels (mmol/L), HbA1c %.

CONTACTS AND LOCATIONS:
Overall Officials: Ran Tian, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] You DG, Saravanakumar G, Son S, Han HS, Heo R, Kim K, Kwon IC, Lee JY, Park JH. Dextran sulfate-coated superparamagnetic iron oxide nanoparticles as a contrast agent for atherosclerosis imaging. Carbohydr Polym. 2014 Jan 30;101:1225-33. doi: 10.1016/j.carbpol.2013.10.068. Epub 2013 Oct 26. PMID 24299895
- [Background] Celermajer DS, Sorensen KE, Gooch VM, Spiegelhalter DJ, Miller OI, Sullivan ID, Lloyd JK, Deanfield JE. Non-invasive detection of endothelial dysfunction in children and adults at risk of atherosclerosis. Lancet. 1992 Nov 7;340(8828):1111-5. doi: 10.1016/0140-6736(92)93147-f. PMID 1359209
- [Background] Tremaroli V, Backhed F. Functional interactions between the gut microbiota and host metabolism. Nature. 2012 Sep 13;489(7415):242-9. doi: 10.1038/nature11552. PMID 22972297
- [Background] Matsuzawa Y, Kwon TG, Lennon RJ, Lerman LO, Lerman A. Prognostic Value of Flow-Mediated Vasodilation in Brachial Artery and Fingertip Artery for Cardiovascular Events: A Systematic Review and Meta-Analysis. J Am Heart Assoc. 2015 Nov 13;4(11):e002270. doi: 10.1161/JAHA.115.002270. PMID 26567372
- [Background] Karlsson FH, Fak F, Nookaew I, Tremaroli V, Fagerberg B, Petranovic D, Backhed F, Nielsen J. Symptomatic atherosclerosis is associated with an altered gut metagenome. Nat Commun. 2012;3:1245. doi: 10.1038/ncomms2266. PMID 23212374
- [Background] Affuso F, Ruvolo A, Micillo F, Sacca L, Fazio S. Effects of a nutraceutical combination (berberine, red yeast rice and policosanols) on lipid levels and endothelial function randomized, double-blind, placebo-controlled study. Nutr Metab Cardiovasc Dis. 2010 Nov;20(9):656-61. doi: 10.1016/j.numecd.2009.05.017. Epub 2009 Aug 20. PMID 19699071
- [Background] Xie W, Gu D, Li J, Cui K, Zhang Y. Effects and action mechanisms of berberine and Rhizoma coptidis on gut microbes and obesity in high-fat diet-fed C57BL/6J mice. PLoS One. 2011;6(9):e24520. doi: 10.1371/journal.pone.0024520. Epub 2011 Sep 6. PMID 21915347
- [Background] Wang Y, Shou JW, Li XY, Zhao ZX, Fu J, He CY, Feng R, Ma C, Wen BY, Guo F, Yang XY, Han YX, Wang LL, Tong Q, You XF, Lin Y, Kong WJ, Si SY, Jiang JD. Berberine-induced bioactive metabolites of the gut microbiota improve energy metabolism. Metabolism. 2017 May;70:72-84. doi: 10.1016/j.metabol.2017.02.003. Epub 2017 Feb 10. PMID 28403947
- [Background] Cao Y, Pan Q, Cai W, Shen F, Chen GY, Xu LM, Fan JG. Modulation of Gut Microbiota by Berberine Improves Steatohepatitis in High-Fat Diet-Fed BALB/C Mice. Arch Iran Med. 2016 Mar;19(3):197-203. PMID 26923892